CLINICAL TRIAL: NCT03212183
Title: Evaluation of a Web-based Virtual Nursing Intervention to Support Self-Management Among Adults With Epilepsy: A Preliminary Study
Brief Title: Evaluation of a Web-based Virtual Nursing Epilepsy Self-Management Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Savoy Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17.136
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2018-01

CONDITIONS: Epilepsy
Keywords: web-based intervention; self-management; nursing; epilepsy; seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPI-TAVIE (Experimental): Patients assigned to this arm will be invited to complete a web-based nursing intervention called EPI-TAVIE.
  Interventions: Behavioral: EPI-TAVIE
- Websites (Other): Patients assigned to this arm will be invited to consult a validated list of predetermined conventional websites.
  Interventions: Other: Websites

INTERVENTIONS:
Behavioral: EPI-TAVIE — ÉPI-TAVIE is a web-based intervention focusing on epilepsy self-management. This interactive session (25 minutes) is facilitated by a virtual nurse.
  Arms: EPI-TAVIE
Other: Websites — The conventional websites offers reliable information about epilepsy. Their content were validated by experts.
  Arms: Websites

SUMMARY:
The purpose of this pilot randomized controlled trial is to evaluate a web-based virtual nursing intervention (ÉPI-TAVIE) in terms of 1) acceptability and feasibility, and; 2) preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* to be a patient of the Clinique d'épilepsie du Centre Hospitalier de l'Université de Montréal
* to be able to read and understand French
* to have access to the Internet

Exclusion Criteria:

* having an uncontrolled psychiatric or cognitive condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

PRIMARY OUTCOMES:
Self-management | 3 months
  Self-management will be measured with the Epilepsy Self-Management Scale (Dilorio et al., 1994). The scale is composed of 38 items that assess the degree to which people perform tasks to manage their epilepsy. It is composed of five subscales: medication management, information management, seizure management, safety management and lifestyle management.

SECONDARY OUTCOMES:
Acceptability of the intervention | 1 month
  Acceptability will be evaluated through a self-administered questionnaire composed of items regarding satisfaction with the approach, convenience of use, ease of understanding, relevance, dosage and overall appreciation (Côté et al., 2012).
Feasibility of the intervention | 1 month
  Feasibility will be assessed by an evaluation of exposition to intervention: for each participants, the number of page viewed will be recorded. Fidelity to the intervention structure will be obtained by comparing the projected number of pages view to the number of viewed pages, thus addressing its feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: José Côté, PhD, Principal Investigator — CRCHUM, Université de Montréal; Dang Khoa Nguyen, PhD, Study Chair — CHUM, Université de Montréal, CRCHUM; Line Beaudet, PhD, Study Chair — CHUM, Université de Montréal, CRCHUM; Yann-Gaël Guéhéneuc, PhD, Study Chair — Polytechnique Montréal; Vanessa Léger, BScN, Study Chair — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cote J, Beaudet L, Auger P, Rouleau G, Chicoine G, Leger V, Keezer M, Reid MA, Nguyen DK. Evaluation of a web-based virtual nursing intervention to support self-management among adults with epilepsy: A mixed-methods study. Epilepsy Behav. 2021 Jan;114(Pt A):107581. doi: 10.1016/j.yebeh.2020.107581. Epub 2020 Nov 25. PMID 33246896